CLINICAL TRIAL: NCT00193024
Title: A Phase II Trial of Epirubicin/Docetaxel in the First-Line Treatment of Patients With Metastatic Breast Cancer
Brief Title: Epirubicin and Docetaxel in the Treatment of Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Pharmacia and Upjohn (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 39; 378-ONC-0030-219; GIA 11168
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin

INTERVENTIONS:
Drug: Docetaxel
Drug: Epirubicin

SUMMARY:
The epirubicin/docetaxel combination is one of the most active and best tolerated taxane/anthracycline combinations. In this phase II trial, we will further evaluate the feasibility, safety and effectiveness of the docetaxel/epirubicin combination, when administered as first-line treatment for metastatic breast cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will receive:

Docetaxel + Epirubicin

Both drugs will be repeated at 21-day intervals

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic breast cancer confirmed by biopsy.
* Received no previous chemotherapy for metastatic breast cancer.
* Prior hormonal therapy is acceptable.
* Measurable or evaluable disease.
* Able to perform activities of daily living without considerable assistance
* Adequate bone marrow, liver and kidney function
* Must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years.
* Cardiac ejection fraction < 45%.
* Women who are pregnant or lactating.
* Patients with meningeal metastases are ineligible.
* Moderate peripheral neuropathy
* History of hypersensitivity reaction to Taxotere
* Males with metastatic breast cancer

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2001-09; Primary Completion 2003-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Clinical response rate of the docetaxel/epirubicin combination in the first-line treatment of patients with metastatic breast cancer

SECONDARY OUTCOMES:
Safety of the docetaxel/epirubicin combination in the first-line treatment of patients with metastatic breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Yardley DA, Spigel DR, Meluch AA, Rinaldi D, Schnell FM, Greco FA. Docetaxel and epirubicin as first-line treatment for patients with metastatic breast cancer: a Minnie Pearl Cancer Research Network Phase II trial. Cancer Invest. 2006 Aug-Sep;24(5):469-73. doi: 10.1080/07357900600814060. PMID 16939953